CLINICAL TRIAL: NCT02694666
Title: Effects of Controlled Whole-body Vibration Training on Preventing Falls Among Healthy Population and Ambulatory People With Multiple Sclerosis
Brief Title: Vibration Training for Preventing Falls in Healthy Population and Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Feng Yang, PhD, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 514810
Record Dates: First submitted 2016-02-10; First posted 2016-02-29 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Falls Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration training group (Experimental): The vibration group will receive 8-week controlled whole-body vibration training as the intervention on the Galileo Med L device
  Interventions: Other: Controlled whole-body vibration training
- Placebo training group (Placebo Comparator): The placebo group will receive 8-week placebo training on the Galileo Med L device
  Interventions: Other: Controlled whole-body vibration training

INTERVENTIONS:
Other: Controlled whole-body vibration training — The intervention is an 8-week program
  Other Names: Vibration therapy; vibration training

SUMMARY:
This study is to investigate the effects of controlled whole-body vibration training on reducing the likelihood of falls among healthy population and people with multiple sclerosis. (NOTE: research not covered by sponsored funding)

DETAILED DESCRIPTION:
For each population, the participants will be randomized into two groups.

ELIGIBILITY:
Inclusion Criteria:

For healthy population:

* Aged between 18 and 75
* No known history of musculoskeletal, neurological, cardiovascular, or pulmonary impairment

For people with multiple sclerosis

* Self-reported multiple sclerosis and confirmed by the physician
* No significant relapse within the past 8 weeks
* To be able to walk independently a length of 25 feet
* Score on Patient Determined Disease Step < 7

Exclusion Criteria:

* Subjects use any sedative of any type.
* The heel bone density is less than -2.0

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-04; Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Real life falls | Up to 12 months
  Real life falls are monitored for 12 months.

SECONDARY OUTCOMES:
Berg Balance Scale test | Up to 12 months
  This test is used to assess the body balance skill in healthy elderly.
Slip-related falls on treadmill | Up to 12 months
  Participants will be exposed to unexpected slips during walking on a treadmill.
Functional mobility | Up to 12 months
  Functional mobility is measured by using the Timed-Up-and-Go test.
Sensation | Up to 12 months
  Sensation is measured by nylon monofilaments kit.
Muscle strength | Up to 12 months
  Lower-limb joints' muscle strengths are evaluated by an isokinetic dynamometer.
Range of motion | Up to 12 months
  The range of motion of the lower limb joints are assessed by a goniometer.
Bone density | Up to 12 months
  The bone density of the heel bone is assessed by a bone ultrasonometer.
Multiple Sclerosis Functional Composite score | Up to 12 months
  The Multiple Sclerosis Functional Composite score, which indicates the disability level in people with multiple sclerosis, is measured
Equiscale balance test | Up to 12 months
  This balance test is applied to individuals with multiple sclerosis to evaluate their body balance skill.
Symbol Digit Modalities test | Up to 12 months
  This test measures participants' attention and information processing speed and efficiency.
Selective Reminding test | Up to 12 months
  This instrument assesses participants' verbal learning and memory capacity.
Behavior Rating Inventory of Executive Function | Up to 12 months
  This test is used to gauge one's everyday behaviors associated with specific domains of the executive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yang, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang F, Su X, Sanchez MC, Hackney ME, Butler AJ. Vibration training reducing falls in community-living older adults: a pilot randomized controlled trial. Aging Clin Exp Res. 2023 Apr;35(4):803-814. doi: 10.1007/s40520-023-02362-6. Epub 2023 Feb 13. PMID 36781617